CLINICAL TRIAL: NCT07168226
Title: A Multi-center, Randomized, Phase 2 Clinical Trial to Exploratively Evaluate the Efficacy and Safety of ASCA101 for the Treatment of Cachexia in Patients With Solid Tumor
Brief Title: Phase 2 Cachexia Clinical Trial to Evaluate the Efficacy and Safety of ASCA101
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MetaFines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MF-ASCA101-03
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ASCA101 Inj. 24.32mg/kg #1 (Experimental): ASCA101 injection 24.32 mg/kg administered twice a week in study 1
  Interventions: Drug: ASCA101 24.32mg/kg
- ASCA101 Inj. 32.43mg/kg #1 (Experimental): ASCA101 injection 32.43 mg/kg administered twice a week in study 1
  Interventions: Drug: ASCA101 32.43mg/kg
- Megace F suspension (Active Comparator): Megace F suspension(20mL) administered daily in study 1
  Interventions: Drug: Active Comparator
- ASCA101 Inj. 24.32mg/kg #2 (Experimental): ASCA101 injection 24.32 mg/kg administered twice a week in study 2
  Interventions: Drug: ASCA101 24.32mg/kg
- ASCA101 Inj. 32.43mg/kg #2 (Experimental): ASCA101 injection 32.43 mg/kg administered twice a week in study 2
  Interventions: Drug: ASCA101 32.43mg/kg
- Placebo (Placebo Comparator): 0.9% normal saline injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Comparator — Megace F suspension 20mL, intake daily for 12weeks
  Arms: Megace F suspension
Drug: ASCA101 24.32mg/kg — ASCA101 Inj. 24.32mg/kg, twice a week for 12 weeks
  Arms: ASCA101 Inj. 24.32mg/kg #1; ASCA101 Inj. 24.32mg/kg #2
Drug: ASCA101 32.43mg/kg — ASCA101 Inj. 32.43mg/kg, twice a week for 12 weeks
  Arms: ASCA101 Inj. 32.43mg/kg #1; ASCA101 Inj. 32.43mg/kg #2
Drug: Placebo — 0.9% normal saline injection
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of ASCA101 for the treatment of Cachexia in solid tumor patients. The main questions it aims to answer are:

Can the efficacy of ASCA101 in improving cachexia be evaluated based on changes in body weight measured by InBody after 12 weeks (3 cycles) of weekly administration, compared to baseline, for each dose group?

Do participants experience adverse events during administration of ASCA101 and/or within 4 weeks after the end of administration?

This clinical trial comprises two parts. [Study 1. Active-Controlled, Open-Label Study] Participants who provide written informed consent will undergo screening procedures. Those who meet all inclusion criteria and none of the exclusion criteria will be eligible for enrollment and will be randomized to receive either ASCA101 (at one of two dose levels: 24.32 or 32.43 mg/kg) or an active control. Participants will receive the investigational product over 3 cycles (12 weeks). Each cycle consists of 28 days. Subjects in the ASCA101 group will receive the investigational drug twice weekly for a total of 8 doses per cycle. Participants in the active control group (megace F suspension) will receive the drug orally once daily.

[Study 2. Placebo-Controlled, Double-Blind Study] Participants who provide written informed consent will undergo screening procedures. Those who meet all inclusion criteria and none of the exclusion criteria will be eligible for enrollment and will be randomized to receive either ASCA101 (at one of two dose levels: 24.32 or 32.43 mg/kg) or placebo. Participants will receive the investigational product over 3 cycles (12 weeks). Each cycle consists of 28 days. Subjects in the ASCA101 group will receive the investigational drug twice weekly for a total of 8 doses per cycle. Participants in the placebo group will receive placebo in the same manner as the ASCA101 group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 years or older with a histologically or cytologically confirmed diagnosis of a solid tumor (primary tumor types: colorectal cancer, ovarian cancer, and lung cancer [lung cancer applicable to Study 1 only]).
2. (For female subjects only): Must be either surgically sterilized or postmenopausal*.

   *Postmenopause is defined as the permanent cessation of ovarian function, evidenced by the absence of menstruation for 12 consecutive months not attributable to other medical causes.
3. Must meet at least one of the following criteria consistent with cachexia diagnosis*:

   ① Unintentional weight loss of >5% over the past 6 months, or

   ② BMI <20 kg/m² with unintentional weight loss of >2% over the past 6 months, or

   ③ Diagnosis of sarcopenia (skeletal muscle index: <7.26 kg/m² for men, <5.45 kg/m² for women) with unintentional weight loss of >2% over the past 6 months.

   *For subjects requiring confirmation of sarcopenia for cachexia diagnosis, skeletal muscle mass must be assessed using Dual-Energy X-ray Absorptiometry (DEXA).
4. Clinical laboratory results measured within 14 days prior to randomization must meet the following criteria (without G-CSF administration or blood transfusion within 14 days prior to lab tests):

   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm³

     * Platelet count ≥ 100,000/mm³ ③ Hemoglobin ≥ 9.0 g/dL

       * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) ⑤ Total bilirubin ≤ 1.5 × ULN ⑥ AST and ALT ≤ 3 × ULN (≤ 5 × ULN if liver metastasis is present) ⑦ INR and aPTT ≤ 1.5 × ULN
5. Able to consume food orally.
6. Able to complete questionnaires.
7. Life expectancy of at least 16 weeks, as assessed by the investigator.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
9. Male subjects who have not undergone vasectomy must agree to use highly effective contraception from at least 4 weeks prior to study drug administration, throughout the study period, and for 6 months following the last dose.

   Highly effective contraception includes: partner's hormonal contraception, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, or total sexual abstinence.
10. Able and willing to voluntarily provide written informed consent to participate in this clinical trial.

Exclusion Criteria:

1. Subjects scheduled to undergo surgery for cancer treatment or currently receiving/planned to receive non-chemotherapy anticancer therapies such as radiotherapy, hormone therapy, or immunotherapy.
2. History of hypersensitivity to any component of the investigational product or to drugs of the same class.
3. Currently taking medications for the purpose of appetite stimulation or weight gain.
4. History of surgery within 6 months prior to screening. (Note: Subjects undergoing postoperative chemotherapy are eligible regardless of the time of surgery.)
5. Subjects requiring dietary restrictions.
6. Subjects requiring enteral or parenteral nutrition.
7. Weight loss due to causes other than malignancy, including:

   * Major endocrine/metabolic disorders (e.g., hyperthyroidism, uncontrolled diabetes mellitus)
   * Conditions affecting appetite or calorie intake (e.g., mechanical bowel obstruction, cholestasis, uncontrolled nausea/vomiting, malabsorption syndromes, severe diarrhea)
8. Conditions that may lead to weight gain, including major endocrine/metabolic diseases (e.g., hypothyroidism, Cushing's syndrome).
9. History of any of the following cardiovascular conditions within the past 5 years:

   * Congestive heart failure (CHF) classified as NYHA Class II or higher, or LVEF

     * 50%
   * Uncontrolled hypertension (SBP/DBP >140/90 mmHg)
   * History of hypertensive crisis or hypertensive encephalopathy
   * Pulmonary hypertension
   * Myocardial infarction
   * Clinically significant vascular disease within 6 months prior to the first dose (e.g., aneurysm requiring surgery, recent peripheral arterial thrombosis)
   * Uncontrolled arrhythmias
10. Persistent clinically significant toxicity (Grade ≥2 per NCI-CTCAE v5.0) due to previous cancer treatment.
11. Subjects with severe infections or severe traumatic systemic conditions.
12. Symptomatic or uncontrolled central nervous system (CNS) metastases. (Note: Subjects with asymptomatic CNS metastases who have discontinued systemic corticosteroids at least 4 weeks prior to randomization and have been radiologically and neurologically stable for ≥4 weeks are eligible.)
13. History of contraindications to ascorbic acid or calcium injections, including:

    * Hyperoxaluria, thalassemia
    * Gout, cystinuria
    * Glucose-6-phosphate dehydrogenase (G6PD) deficiency
    * History of kidney stones with hypercalciuria
    * Hypercalcemia (Ca ≥10.5 mg/dL)
    * Sarcoidosis
    * Nephrolithiasis
    * Hypoproteinemia (Total protein ≤6.0 g/dL)
    * Severe renal impairment (eGFR < 30 mL/min)
14. Patients with severe neurological or psychiatric disorders that, in the investigator's judgment, are sufficient to affect the clinical trial outcomes (e.g., depression, dementia, delirium).
15. Patients who are breastfeeding or who, or whose partners, are planning to become pregnant during the clinical trial period.
16. Individuals who have participated in another clinical trial within 30 days prior to screening.
17. Patients with a history of bleeding-related or gastrointestinal diseases, as described below:

    * Evidence of active bleeding, bleeding diathesis, coagulopathy, or tumors involving major blood vessels.
    * Clinically significant peptic ulcers, gastrointestinal bleeding, gastrointestinal or non-gastrointestinal fistulas, perforations, intra-abdominal abscesses, signs or symptoms of gastrointestinal obstruction, requirement of parenteral hydration or nutrition, or a history of inflammatory bowel disease (IBD).
    * Evidence of free air in the abdomen not explained by paracentesis or recent surgical procedures.
18. Patients who have received biguanides (e.g., metformin) within 2 weeks prior to screening or are expected to require them during the clinical trial.
19. Patients requiring continuous systemic corticosteroid therapy (exceptions allowed as below):

    * Use of local corticosteroids such as intra-articular, intranasal, ophthalmic, or inhaled corticosteroids is permitted.
    * Temporary systemic corticosteroid use for treatment or prevention of contrast agent allergy or adverse events is allowed.
20. Patients with HIV or other severe diseases deemed by the investigator to make study participation inappropriate.
21. Patients who underwent drainage of ascites and/or pleural effusion within 14 days prior to screening.
22. Patients with hemoptysis (defined as ≥1/2 teaspoon of bright red blood per episode) within 14 days prior to screening.
23. Patients who underwent core biopsy or other minor surgical procedures (excluding vascular access device placement) within 14 days prior to the first administration of the investigational product.
24. Patients with significant, unhealed wounds, active ulcers, or untreated fractures.
25. Patients with a history of cerebrovascular accident (stroke), transient ischemic attack, or subarachnoid hemorrhage within 6 months prior to screening.
26. Patients with a history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
27. Any other condition deemed by the investigator to make the patient unsuitable for participation in the clinical trial.

    [Exclusion Criteria Applicable Only to Study 1]
28. Patients with a history of hypersensitivity to megestrol acetate or any of its components.
29. Patients with a history of thromboembolic disease.
30. Patients with diabetes mellitus.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight at the end of cycle 3 compared to baseline | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days.)
  Change in body weight measured by InBody at the end of cycle 3 compared to baseline

SECONDARY OUTCOMES:
Change in body weight at the end of cycle 1 & cycle 2 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2. (Each cycle is 28days)
  Change in body weight measured by InBody at the end of cycle 1 & cycle 2 compared to baseline
Percentage of subjects with ≥5% increase in body weight at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Percentage of subjects with ≥5% increase in body weight measured by InBody at the end of cycle 1, cycle 2 and cycle 3 compared to baseline
Change in body weight at the end of cycle 1, cycle 2 and cycle 3 compared to baseline measured by DEXA | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in body weight(unit: kilograms) measured by DEXA(Dual-Energy X-ray Absorptiometry) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline.
Change in appendicular skeletal muscle mass (ASM) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline measured by DEXA | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in ASM (unit: kilograms) measured by DEXA (Dual-Energy X-ray Absorptiometry) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline. ASM is calculated by summing the lean soft tissue mass of the arms and legs (appendicular regions) measured by DEXA.
Change in appendicular bone mineral content at the end of cycle 1, cycle 2 and cycle 3 compared to baseline measured by DEXA | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in appendicular bone mineral content(unit: grams or kilograms) measured by DEXA(Dual-Energy X-ray Absorptiometry) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline. It is calculated by measuring the bone mineral content (BMC) of the arms and legs using DEXA and then summing the values.
Change in appendicular skeletal muscle mass index (ASMI) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline measured by DEXA | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in ASMI (unit: kg/m²) measured by DEXA(Dual-Energy X-ray Absorptiometry) at the end of cycle 1, cycle 2 and cycle 3 compared to baseline. It is calculated by dividing ASM (kg) by height squared (m²).
Change in lean body mass and fat mass at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in lean body mass and fat mass (unit: kilograms) measured by InBody and DEXA the end of cycle 1, cycle 2 and cycle 3 compared to baseline.
Change in skeletal muscle mass and lower limb muscle mass at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in skeletal muscle mass and lower limb muscle mass measured by InBody at the end of cycle 1, cycle 2 and cycle 3 compared to baseline.
Change in Timed Up and Go test (TUG) results at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3 (each cycle is 28days)
  The Timed Up and Go (TUG) test is performed with the patient starting in a seated position. Upon a signal, the patient stands up, walks approximately 3 meters (10 feet), turns around, and returns to sit in the chair. The time taken (in seconds) to complete this task is measured. Completion within 10 seconds is considered normal, and longer times are interpreted as indicating reduced mobility and increased risk of falls.
Change in PGIC-C and PGIC-S at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Both PGIC-C and PGIC-S are patient-reported outcome (PRO) measures used to directly assess the patient's perceived change in condition following treatment. PGIC-C (Patient Global Impression of Change - Condition) evaluates the patient's overall change in condition using a 7-point Likert scale, with scores of 1-2 indicating marked improvement and scores of 5-7 indicating worsening. PGIC-S (Patient Global Impression of Change - Symptoms) assesses the patient's perceived change in specific symptoms, also using a 7-point Likert scale, with scores of 1-2 indicating marked improvement in symptoms and scores of 5-7 indicating worsening of symptoms.
Change in FAACT - Appetite domain score at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. (Each cycle is 28days)
  Change in FAACT(Functional Assessment of Anorexia/Cachexia Therapy) - Appetite domain score at the end of cycle 1, cycle 2 and cycle 3 compared to baseline. FAACT - Appetite domain score is a patient-reported outcome (PRO) measure used to assess the patient's appetite. Each item is rated on a 5-point Likert scale, and the domain score is calculated by summing the item scores. Higher scores indicate better appetite and lower symptom severity.
Change in FACIT-F score at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3 (each cycle is 28days)
  FACIT-F (Functional Assessment of Chronic Illness Therapy - Fatigue) score is a patient-reported outcome (PRO) measure used to assess the level of fatigue in patients with chronic illnesses. It consists of 13 items, each rated on a 0-4 Likert scale. The total score is calculated by summing the item scores, with higher scores indicating less fatigue and better overall condition.
Change in handgrip strength at the end of cycle 1, cycle 2 and cycle 3 compared to baseline | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3 (each cycle is 28days)
  Handgrip strength is assessed using a digital or spring dynamometer, with the patient seated, elbow flexed at 90°, and wrist in a neutral position. Each hand is measured 1-3 times, and the maximum value is recorded. Grip strength criteria (kg) vary by sex and age group, and values below the reference are considered indicative of low muscle strength.

OTHER OUTCOMES:
Exploratory outcome : Adverse Events | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  Adverse events will be summarized by treatment group, including overall adverse events (TEAEs), adverse drug reactions (ADRs), serious adverse events (SAEs), and adverse events leading to study discontinuation. For each category, the frequency, percentage, number of occurrences, and incidence rate will be presented along with two-sided 95% confidence intervals.
Clinical laboratory tests : Hematology Tests | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  To conduct Hematology Tests, blood samples are analyzed using an automated hematology analyzer. Parameters of the tests are White blood cells (WBC), red blood cells (RBC), hemoglobin (Hb), platelets (PLT), etc.
Clinical laboratory tests : Blood Chemistry Tests | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  To conduct Blood Chemistry Tests, using automated chemistry analyzer or immunoassay. Parameters of the tests are liver function (ALT, AST), kidney function (Creatinine, BUN), electrolytes (Na, K, Cl), glucose, lipids, etc.
Clinical laboratory tests : Coagulation Tests | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  To conduct Coagulation Tests, plasma samples analyzed using an automated coagulation analyzer. PT (Prothrombin Time), aPTT (Activated Partial Thromboplastin Time), INR.
Clinical laboratory tests : Urinalysis | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  To conduct Urinalysis, using reagent strips or an automated urine analyzer. Parameters of the test are color, specific gravity, pH, protein, glucose, red/white blood cells, ketones, etc.
Vital signs : Blood pressure | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cyle is 28days.
  Vital signs should be assessed prior to any planned procedures whenever possible, after the subject has rested in a seated position. Blood pressure measured in the seated position using an automated sphygmomanometer with an appropriately sized cuff. At least two readings will be obtained, separated by 1-2 minutes, and the average will be recorded. The unit of measurement for blood pressure is millimeters of mercury (mmHg).
Vital signs : Pulse | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cyle is 28days.
  Pulse is measured simultaneously with blood pressure using the automated device, or manually by radial palpation for 30 seconds and extrapolated to beats per minute (bpm).
Vital signs : Body temperature | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cyle is 28days.
  Body temperature is measured using a calibrated digital thermometer, preferably via the oral or tympanic route, and recorded in degrees Celsius (°C).
Exploratory outcome : Physical examination | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  At each visit, a physical examination will be performed, including inspection, palpation, percussion, and auscultation, to assess the subject's overall health and to identify any adverse events. The physical examination will include evaluation of the general appearance, skin, head/neck, chest/lungs, heart, abdomen, genitourinary system, extremities, musculoskeletal system, nervous system, and lymph nodes.
Electrocardiogram (ECG) : PR interval, QRS interval, QT interval and QTc interval | At Screening, baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3, EOS (4 weeks after end of cycle 3). Each cycle is 28days.
  PR interval, QRS interval, QT interval and QTc interval will be measured by ECG. All of them are expressed in milliseconds (ms). The PR interval, which measures the conduction time from the atria to the ventricles, has a normal range of 120-200 ms. The QRS complex, representing the duration and width of ventricular depolarization, has a normal range of 80-120 ms. The QT interval, representing the duration of ventricular depolarization and repolarization, can also be reported in its corrected form (QTc).
Central lab assessments: GDF-15 | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. Each cycle is 28days.
  Blood samples for central laboratory testing will be obtained after an overnight fast of at least 8 hours, prior to administration of the investigational medicinal product. Water intake is permitted during the fasting period. Samples will be collected in serum or plasma tubes, processed by centrifugation, stored at -80 °C, and shipped to the central laboratory for analysis.
  GDF-15 results are expressed in pg/mL. Elevated levels are associated with aging, cardiovascular disease, cancer, and cachexia.
Central lab assessments: Interleukin-1β (IL-1β) | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. Each cycle is 28days.
  Blood samples for central laboratory testing will be obtained after an overnight fast of at least 8 hours, prior to administration of the investigational medicinal product. Water intake is permitted during the fasting period. Samples will be collected in serum or plasma tubes, processed by centrifugation, stored at -80 °C, and shipped to the central laboratory for analysis.
  Interleukin-1β results are expressed in pg/mL. Detectable levels above baseline indicate systemic or local inflammatory activity.
Central lab assessments: Interleukin-6 (IL-6) | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. Each cycle is 28days.
  Blood samples for central laboratory testing will be obtained after an overnight fast of at least 8 hours, prior to administration of the investigational medicinal product. Water intake is permitted during the fasting period. Samples will be collected in serum or plasma tubes, processed by centrifugation, stored at -80 °C, and shipped to the central laboratory for analysis.
  Interleukin-6 measured using ELISA or electrochemiluminescence-based methods. Results are expressed in pg/mL. Increased concentrations reflect systemic inflammation, infection, or metabolic dysregulation.
Central lab assessments: Tumor Necrosis Factor-α (TNF-α) | At baseline(0 week), End of Cycle 1, End of Cycle 2, End of Cycle 3. Each cycle is 28days.
  Blood samples for central laboratory testing will be obtained after an overnight fast of at least 8 hours, prior to administration of the investigational medicinal product. Water intake is permitted during the fasting period. Samples will be collected in serum or plasma tubes, processed by centrifugation, stored at -80 °C, and shipped to the central laboratory for analysis.
  TNF-α quantified by ELISA or multiplex cytokine assay. Results are expressed in pg/mL. Elevated levels are associated with chronic inflammation, autoimmune disorders, and metabolic diseases.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Gyeonggi-do, Goyang-si
  - Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do, Gwangmyeong-si
  - Seoul ST. Mary's hospital, Seoul, Seocho-gu
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - Ajou University Hospital, Gyeonggi-do, Suwon-si